CLINICAL TRIAL: NCT06981416
Title: The Effect of Digital and Classical Education Based on Planned Behavior Theory Given to Mothers in the Risk Group on Their Self-Efficacy in Identifying Safety Measures and First Aid for Home Accidents: A Randomized Controlled Trial
Brief Title: The Effect of Digital and Classical Education Based on Planned Behavior Theory Given to Mothers in the Risk Group on Their Self-Efficacy in Identifying Safety Measures and First Aid for Home Accidents
Acronym: Home Accidents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SU-2025
Record Dates: First submitted 2025-04-21; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Nursing
Keywords: Drowning, Child, Fall, Electric Shock, Home accidents, First Aid, Burn, Poisoning,
MeSH Terms: conditions — Drowning; Burns; Poisoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group (Dijital education) (Experimental): The mothers in this group will be given an educational animation video based on the "Planned Behavior Theory" as a single session asl digital training.
  Interventions: Behavioral: Digital education group
- intervention group (classical education) (Experimental): The mothers in this group will receive classical education in the form of a flow chart, with educational content prepared according to the "Planned Behavior Theory".
  Interventions: Behavioral: classical education group
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Digital education group — Digital training for home accidents and first aid based on the Theory of Planned Behavior (PBT) and the pre-test, post-test and follow-up results will be evaluated.
  Other Names: intervention1
  Arms: intervention group (Dijital education)
Behavioral: classical education group — The training content prepared according to the "Planned Behavior Theory" will be given as classical training in the form of a flow chart.
  Other Names: intervention2
  Arms: intervention group (classical education)

SUMMARY:
Childhood home accidents are a significant health problem in our country and the world. Home accidents are more common in children aged 1-5, and cause temporary and permanent disabilities in deaths.

In the project proposal, it is planned to conduct a randomized controlled trial to determine the effects of digital and classical home accident and first aid training given to mothers in the risk group with children aged 1-3 in line with the Planned Behavior Theory (PDT) on home accident safety precautions and first aid self-efficacy.

In the study, the features of the education model that will provide original value and original contribution are that it is digitally based (animated video) education, which will allow individuals to receive training at their own pace and in accordance with their needs due to its individualizable feature. This will encourage mothers to participate more at the appropriate time and actively participate in the training. It is a more cost-effective and time-saving application compared to other teaching materials. In addition, it is original in that the group to be trained is mothers in the risk group. It is different from other studies on 'home accidents' in that it is planned in line with the PDT, randomized controlled, and the outputs will be measured with repeated measurements.

The implementation of this project will consist of four main stages. In the first stage, the creation of the educational content, preparation of digital and classical educational materials in line with expert opinions and their evaluation by expert opinions. In the second stage, the final version will be arranged in line with the preliminary application. In the third stage, the implementation of the initiative and the collection of data. In the fourth stage, the statistical analysis of the data.

The total duration of the project will be divided into approximately 3 months in the first stage, 1 month in the second, 7 months in the third and the last stage in the 1-month stage. In order for the project to be carried out healthily and effectively, the project manager and the doctoral student specialist nurse will take part.

Since the project is original, if it is successful, there is a high probability that a doctoral thesis will be formed. It is highly likely that a researcher with a doctorate title will be formed upon completion of the project. The importance of the digital education method is very clear and its active use in nursing education will positively contribute to the development of child and family health. It is highly probable that the training model to be created will be recommended for use in secondary and tertiary healthcare institutions, including primary healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Being a mother with a 1-3 year old child,
* Having a low socioeconomic status (income below the poverty line) https://www.who.int/data/gho/indicator-metadata-registry/imr-details/4744 ,
* Being the primary caregiver is the mother,
* The mother is literate,
* The mother is willing to participate in the study.

Exclusion Criteria:

* The child has a mental or physical disability,
* The mother is a health worker,
* The mother has been diagnosed with a mental or psychiatric illness

Max Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Mothers will be included in the study.
Enrollment: 108 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Scale for Identifying Mothers' Safety Measures Against Home Accidents in 6-Year-Old Children | before the educational (pre-test), after the educational (post-test) and after the education 3 months (follow-up)
  The scale was developed by Çınar and Görak (2003). The scale defines the precautions taken by mothers with children between the ages of 0-6 to protect themselves from home accidents. The scale consists of 40 items, 34 of which are positively expressed and 6 of which are negatively expressed. The scale is a five-point Likert-type scale, with 34 questions containing positive expressions being scored as always 5 points, often 4 points, sometimes 3 points, rarely 2 points, and never 1 point. Propositions containing negative expressions are items 6, 9, 23, 26, 30, and 40, and the scoring is done in reverse. The minimum scale score is 40, and the maximum scale score is 200 points. As the score obtained from the scale increases, the level of precautions taken by parents increases. The Croncbach alpha internal consistency coefficient value is 0.82
Self-Efficacy of First Aid Scale for Home Accidents | before the educational (pre-test), after the educational (post-test) and after the education 3 months (follow-up)
  he original scale name is "Self-Efficacy of First Aid Scale For Home Accidents" and was developed by Wei and colleagues in 2013 (Wei et al 2013). The scale was adapted to Turkish by Altundağ, Turan and Şafak (2020). The Self-Efficacy of First Aid Scale for Home Accidents consists of 12 items that include interventions that the mother can implement in the event of home accidents. The scale expressions are five-point Likert-type and are indicated as completely agree (100%), completely disagree (0). Higher scores indicate better self-efficacy in first aid. The Cronbach's alpha value of the scale was found to be 0.89

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No